CLINICAL TRIAL: NCT06896734
Title: Evaluation of the mobiCARE™ ECG Monitoring System Electrode Placement Positioning Limits in a Prospective, Non-Randomized, Single-Center U.S. Study
Brief Title: mobiCARE™ ECG Monitoring System
Acronym: SEERS
Status: Completed | Type: Observational
Sponsor: Seers Technology Co., Ltd. (Industry)
Collaborators: Eminence Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEER-CLIN-2024-01
Record Dates: First submitted 2025-02-28; First posted 2025-03-26 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: ECG Monitoring
Keywords: ECG; Heart Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population will include adults who are asymptomatic or who may suffer from transient sympt: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Interventions: Device: Evaluation of the ECG signal in the nominal location and in three alternate positions

INTERVENTIONS:
Device: Evaluation of the ECG signal in the nominal location and in three alternate positions — Evaluation of the ECG signal in the nominal location and in three alternate positions to determine if the three alternate positions are interpretable.

SUMMARY:
Evaluation of the mobiCARE™ ECG Monitoring System Electrode Placement Positioning Limits in a Prospective, Non-Randomized, Single-Center U.S. Study

DETAILED DESCRIPTION:
The purpose of the Seers Technology Company Ltd. sponsored study using the mobiCARE™ ECG Monitoring System is to document the variability and interpretability of heart rhythm tracings from the nominal position whereby the mobiCARE™ device is still able to obtain interpretable ECG signals, in a cohort of adults representative of the U.S. population.

Informational data will be collected, such as P-wave amplitude and QRS amplitude and duration to note any morphological ECG signal changes. Human factors (HF) endpoints will be evaluated including: HCP placement according to IFU, subject demonstration of changing electrodes, dexterity for user to perform the task, electrode placement according to skin markings, and the ability of the user to remove and replace the mobiCARE™ device.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults ≥ 18 years of age;
2. Willing and able to provide informed consent;
3. Able to speak and read English fluently;
4. Participant is ambulatory.

Exclusion Criteria:

1. Patients with cardiac pacemaker;
2. Patients with cardioverter defibrillator;
3. Patients with other implantable electric devices;
4. Currently or has a medical history of skin cancer, rash, skin disorder, keloid, and/or any injury in the chest area;
5. Patients with symptomatic episodes where variations in cardiac performance could result in immediate danger to the patient;
6. Patients with known history of life-threatening arrhythmias;
7. Use in combination with external cardiac defibrillators or high frequency surgical equipment near strong magnetic fields or devices such as MRI;
8. Patients with neuro-stimulator, as it may disrupt the quality of ECG data;
9. Critical care patients;
10. Chest pain at the time of presentation for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MCB Clinical Research Centers, LLC, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim C, Kim SH, Suh MR. Accuracy and Validity of Commercial Smart Bands for Heart Rate Measurements During Cardiopulmonary Exercise Test. Ann Rehabil Med. 2022 Aug;46(4):209-218. doi: 10.5535/arm.22050. Epub 2022 Aug 31. PMID 36071003
- [Background] Rosol M, Petelczyc M, Gasior JS, Mlynczak M. Prediction of peak oxygen consumption using cardiorespiratory parameters from warmup and submaximal stage of treadmill cardiopulmonary exercise test. PLoS One. 2024 Jan 10;19(1):e0291706. doi: 10.1371/journal.pone.0291706. eCollection 2024. PMID 38198496
- [Background] The Prediction of oxygen consumption during Cardiopulmonary exercise test using Wearable ECG (54th Annual Meeting of the Korean Society of Cardiovascular and Thoracic Surgeons 2022 (Alpensia Resort, Pyeongchang, Korea), 2022.11.03-05
- [Background] Kwon S, Choi EK, Lee SR, Oh S, Song HS, Lee YS, Han SJ, Lim HE. Comparison of Novel Telemonitoring System Using the Single-lead Electrocardiogram Patch With Conventional Telemetry System. Korean Circ J. 2024 Mar;54(3):140-153. doi: 10.4070/kcj.2023.0252. PMID 38506104
- [Background] Lee KH, Kim YR, Yoon NS et al. Prediction of Atrial Fibrillation with Single-Lead Mobile ECG during Normal Sinus Rhythm using Deep Learning. e-Cardiology/Digital Health, Public Health, Health Economics, Research Methodology - e-Cardiology/Digital Health, Artificial Intelligence (Machine Learning, Deep Learning. 2024;26 (Supplement 1).
- [Background] Ahn HJ, Choi EK, Lee SR, Kwon S, Song HS, Lee YS, Oh S. Three-Day Monitoring of Adhesive Single-Lead Electrocardiogram Patch for Premature Ventricular Complex: Prospective Study for Diagnosis Validation and Evaluation of Burden Fluctuation. J Med Internet Res. 2024 Mar 21;26:e46098. doi: 10.2196/46098. PMID 38512332
- [Background] Lee HA, Yu W, Choi JD, Lee YS, Park JW, Jung YJ, Sheen SS, Jung J, Haam S, Kim SH, Park JE. Development of Machine Learning Model for VO2max Estimation Using a Patch-Type Single-Lead ECG Monitoring Device in Lung Resection Candidates. Healthcare (Basel). 2023 Oct 30;11(21):2863. doi: 10.3390/healthcare11212863. PMID 37958007
- [Background] Kwon S, Lee SR, Choi EK, Ahn HJ, Song HS, Lee YS, Oh S, Lip GYH. Comparison Between the 24-hour Holter Test and 72-hour Single-Lead Electrocardiogram Monitoring With an Adhesive Patch-Type Device for Atrial Fibrillation Detection: Prospective Cohort Study. J Med Internet Res. 2022 May 9;24(5):e37970. doi: 10.2196/37970. PMID 35532989
- [Background] Kwon S, Lee SR, Choi EK, Ahn HJ, Song HS, Lee YS, Oh S. Validation of Adhesive Single-Lead ECG Device Compared with Holter Monitoring among Non-Atrial Fibrillation Patients. Sensors (Basel). 2021 Apr 30;21(9):3122. doi: 10.3390/s21093122. PMID 33946269
- [Background] Walsh JA 3rd, Topol EJ, Steinhubl SR. Novel wireless devices for cardiac monitoring. Circulation. 2014 Aug 12;130(7):573-81. doi: 10.1161/CIRCULATIONAHA.114.009024. No abstract available. PMID 25114186

RESULTS

PARTICIPANT FLOW:
Groups:
- mobiCARE™ ECG Monitoring System Subjects: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Evaluation of the ECG signal in the nominal location and in three alternate positions: Evaluation of the ECG signal in the nominal location and in three alternate positions to determine if the three alternate positions are interpretable.
Period: Overall Study
Arm/Group | mobiCARE™ ECG Monitoring System Subjects
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Study Population Will Include Adults Who Are Asymptomatic or Who May Suffer From Transient Sympt
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ Ethnicity: Caucasian / non-Hispanic | 26
  Race/ Ethnicity: African American | 8
  Race/ Ethnicity: Asian / Pacific Islander | 2
  Race/ Ethnicity: Hispanic | 9
  Race/ Ethnicity: Native American/Native Alaskan | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Which the ECG Signal is Interpretable at the Nominal Location and up to 3 Alternate Positions
Description: Evaluation of the ECG signal at the nominal location and in up to three (3) additional alternate positions (AP) in each subject to determine if the signal is interpretable. The term "interpretable" is defined as follows: An independent cardiologist reader is able to identify the ECG rhythm in each location when compared to the ECG rhythm measured in the nominal position of the mobiCARE™ Cardiac Monitoring System described in the Instructions for Use. ECG rhythm data will be collected for up to two (2) minutes while the patient ambulates.
  ECG rhythm data were collected in each location during normal use for at least two (2) minutes while the subject was sitting, standing, and ambulating.
  The simultaneous Holter Monitor will be measured at the same time points to have a point of reference for the mobiCARE™ system in the case that changes in the rhythm are noted on the mobiCARE™ Cardiac Monitoring System during the study.
Time Frame: 2 minutes while the patient ambulates
Population: Primary Effectiveness Evaluation: Difference in Interpretability of ECG Signal for MobiCARE™ Nominal and Three Alternative Electrode Placement Locations
Measure: Count of Participants; unit: Participants
Groups:
- Nominal Location: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Evaluation of the ECG signal in the nominal location: Evaluation of the ECG signal in the nominal location to determine if the three alternate positions are interpretable.
- Alternate Position 1: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Evaluation of the ECG signal in the alternate position 1 location: Evaluation of the ECG signal in the alternate position 1 to determine if the three alternate positions are interpretable.
- Alternate Position 2: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Evaluation of the ECG signal in the alternate position 2 location: Evaluation of the ECG signal in the alternate position 2 to determine if the three alternate positions are interpretable.
- Alternate Position 3: The study population will include adults who are asymptomatic or who may suffer from transient symptoms such as arrhythmias and/or palpitations, shortness of breath, dizziness, light headedness, pre-syncope, syncope, fatigue, chest pain and/or anxiety; ranging in age, ethnic group, BMI, educational level and gender.
  Evaluation of the ECG signal in the alternate position 3 location: Evaluation of the ECG signal in the alternate position 3 to determine if the three alternate positions are interpretable.
Arm/Group | Nominal Location | Alternate Position 1 | Alternate Position 2 | Alternate Position 3
Number analyzed (Participants) | 49 | 49 | 49 | 49
Participants | 49 | 49 | 49 | 49

2. Secondary Outcome: Presence of Artifact Graded
Description: Presence of artifact graded as 1=none, 2=minor (cardiac rhythm is interpretable), or 3=major (cardiac rhythm is not interpretable by the independent cardiologist).
Time Frame: 2 minutes
Population: Artifact was rated by the independent ECG reader and rated as 0, 1, or 2. To reflect a more detailed assessment, category 1 was divided into two scores, 1A and 1B. The artifact was categorized according to the definitions below:
  0 = None to negligible artifact
  1A = Minor amount of artifact (≤50% of ECG has artifact); ECG is interpretable
  1. B = Major amount of artifact (>50% of ECG has artifact); ECG is interpretable
  2. = Major (>50% of ECG has artifact); ECG is NOT interpretable.
Measure: Count of Participants; unit: Participants
Groups:
- Nominal Location: Presence of artifact grading at the nominal location
- Alternate Position 1: Presence of artifact grading at alternate position 1
- Alternate Position 2: Presence of artifact grading at alternate position 2
- Alternate Position 3: Presence of artifact grading at alternate position 3
Arm/Group | Nominal Location | Alternate Position 1 | Alternate Position 2 | Alternate Position 3
Number analyzed (Participants) | 49 | 49 | 49 | 49
Participants
  None = 0 - None to negligible artifact | 35 | 21 | 28 | 31
  1A Minor - Minor amount of artifact (≤50% of ECG has artifact); ECG is interpretable | 9 | 14 | 11 | 11
  1B Major - Major amount of artifact (>50% of ECG has artifact); ECG is interpretable | 5 | 14 | 10 | 7
  2 Major - = Major (>50% of ECG has artifact); ECG is NOT interpretable. | 0 | 0 | 0 | 0

3. Secondary Outcome: Evaluation of the ECG Morphology Measurements at the Nominal Position and up to 3 Alternate Positions
Description: The number of measurable positions for QRS amplitude and QRS duration at the nominal position and up to 3 alternate positions.
Time Frame: 2 Minutes
Population: All 49 subjects had measurable QRS complexes in the nominal position and in all three alternate positions, AP #1, AP #2, and AP #3.
Measure: Count of Participants; unit: Participants
Groups:
- Nominal Position; Alternate Position 1; Alternate Position 2; Alternate Position 3: The number of measurable positions for QRS amplitude and QRS duration
Arm/Group | Nominal Position | Alternate Position 1 | Alternate Position 2 | Alternate Position 3
Number analyzed (Participants) | 49 | 49 | 49 | 49
Participants | 49 | 49 | 49 | 49

4. Secondary Outcome: Human Factors Evaluation Measures
Description: Usability Performance Evaluation for Health Care Professionals and Subjects
Time Frame: 2 Minutes
Population: 15 subjects were planned for human factors data collection. 49 subjects were observed for collection of human factors data. The scores for each assessment range from 1 (Difficult) to 5 (Easy). The Healthcare Professional (HCP) and Subject usabilty results are summarized below by mean and standard deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Limited Human Factors Evaluation Measures: Healthcare Professional and Subject Usability
Arm/Group | Limited Human Factors Evaluation Measures
Number analyzed (Participants) | 49
units on a scale
  How easy/difficult for the HCP to place device/electrodes in the Nominal Location using the IFU? | 3.94 (0.92)
  Could the HCP read the ECG signal on app to confirm Lead II/clear signal after the device placed? | 4.43 (0.74)
  How easy/difficult for subject to remove the device/electrodes from Alternate location 3? | 4.1 (1.01)
  How easy or difficult was it for the subject to remove the used electrodes from the mobiCARE™? | 3.67 (1.13)
  How easy/difficult for subject to replace electrodes with new electrodes on the mobiCARE™ device? | 3.69 (1.29)
  How easy or difficult was it for the subject to locate the markings for the nominal position? | 3.49 (1.23)
  How easy/difficult for subject to replace new mobiCARE™ device (electrodes) in the Nominal position | 3.78 (1.23)

5. Secondary Outcome: The Number of Measurable Positions for P-waves
Description: Informational data collected to evaluate interpretability based on P-wave amplitude
Time Frame: 2 minutes
Population: 48 subjects in normal sinus rhythm with measurable P-waves. One subject didn't have a measurable P-wave due to atrial fibrillation. Data is consistent as reported with 48/49 subjects having measurable P-waves.
Measure: Count of Participants; unit: Participants
Groups:
- Nominal Position; Alternate Position 1; Alternate Position 2; Alternate Position 3: The number of measurable positions for P-waves
Arm/Group | Nominal Position | Alternate Position 1 | Alternate Position 2 | Alternate Position 3
Number analyzed (Participants) | 49 | 49 | 49 | 49
Participants | 48 | 48 | 48 | 48

ADVERSE EVENTS:
Time Frame: 2 Minutes
Description: The occurrence and severity of AEs were to be recorded, the occurrence of SAEs was to be recorded, and the occurrence of UADEs was to be recorded in the study.
Groups:
- Adverse Events: Anticipated adverse events observed
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT06896734/Prot_SAP_000.pdf